CLINICAL TRIAL: NCT06309342
Title: Prevention of Lifestyle-related Disorders With Early Examinations of Health and Function and Individualised Functional Profiles - a Randomised Controlled Trial
Brief Title: Prevention of Lifestyle-related Disorders Based on Functional Examinations
Acronym: PREVFUNKTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lena Bornhoft (Other)
Collaborators: Vastra Gotaland Region (Other Government); Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Lena Bornhoft, Research and development leader, Göteborg University
Organization: Göteborg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VGRFOU-278257
Record Dates: First submitted 2024-02-29; First posted 2024-03-13 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Lifestyle-related Condition
Keywords: Lifestyle; Prevention; Physical activity; Fitness; Health examination
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: Initial examinations and data collection are made before randomisation. Randomisation then leads to the two groups of participants receiving different amounts of feedback and support. Follow-up examinations and data collection are made after one year in both groups.
Who Masked: Investigator
Masking Description: Investigators performing the health and function examinations will not be informed about the group to which the participant is allocated. All examinations are performed identically for participants from both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREVFUNKTION (Experimental): Medical examination. Functional examination. Measurement of physical activity. Questionnaires on health, function and lifestyle. Feedback and advice based on medical examination. Feedback and advice based on functional examination. Functional profile. Support in setting goals for lifestyle changes.
  Interventions: Other: PREVFUNKTION; Other: Control
- Control (Active Comparator): Medical examination. Functional examination. Measurement of physical activity. Questionnaires on health, function and lifestyle. Feedback and advice based on medical examination.
  Interventions: Other: Control

INTERVENTIONS:
Other: PREVFUNKTION — Functional profile and advice concerning cardiovascular fitness level, strength, mobility, balance and posture. Motivational interview and support in goalsetting to make lifestyle changes.
  Arms: PREVFUNKTION
Other: Control — Physical activity measured with accelerometers. Functional examination. Medical examination and advice concerning weight measures, blood pressure and standard blood tests.

SUMMARY:
The goal of this randomised controlled trial is to examine the effects of functional examinations and feedback/support on healthy 40-year-olds. The main questions it aims to answer are: • Does feedback and motivational interviewing after testing physical function motivate inactive middle-aged people to increase their physical activity level? • Does the intervention lead to health benefits over time - less pain, better function, higher health-related quality of life, fewer risk factors for lifestyle-related illness? Participants will: • undergo medical and functional health examinations, • their physical activity level will be measured, • receive feedback and advice based on both parts of the examinations, • receive a functional profile, • be supported in goalsetting for lifestyle changes. Researchers will compare with a control group who, after the examinations, receive feedback only from the medical examination to see if participants become more physically active, achieve better function, become more motivated to make lifestyle changes, reduce risk factors for lifestyle-related illness, achieve health benefits and better health-related quality of life.

DETAILED DESCRIPTION:
Relatively healthy 40-year-olds will be examined at baseline and 1 year with both standard medical and newly developed functional examinations and physical activity level will be measured with accelerometers. The intervention group will receive feedback on all their results. A functional profile will be compiled and explained to each participant and they will receive support in setting relevant goals for lifestyle changes and making realistic plans to achieve them. The control group will also be examined as above but will receive feedback and advice based only on the standard medical examination.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age
* Relatively normal general mobility - can walk without support and have no self-reported difficulties with using all four extremities - in order to be able to perform standardised functional performance tests.
* Self-assessed as physically inactive (level 1 or 2 on the Saltin Grimby Physical Activity Level Scale) as inactive people stand to gain most from this intervention.

Exclusion Criteria:

* Verbally self-reported physical activity at level three or four on Saltin Grimby Physical Activity Level Scale.
* Severe mental illness or intellectual impairment, as participants will be expected to fill out questionnaires and should have the ability to follow healthcare advice independently should they choose to do so.
* Pregnancy and/or on-going treatment requiring hospital-based services, to increase probability of baseline values which reflect usual capacity.
* No language restrictions are planned but participants needing interpreter help should arrange this themselves.

Ages: 39 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in objectively measured physical activity | Change between baseline and 1-year follow-up
  Mean daily minutes in moderate-to-very vigorous physical activity measured with accelerometers for 1 week
Change in objectively measured sedentary behaviour | Change between baseline and 1-year follow-up
  Mean daily minutes of sedentary behaviour measured with accelerometers for 1 week

SECONDARY OUTCOMES:
Change in cardiovascular fitness | Change between baseline and 1-year follow-up
  Fitness level measured in ml/kg/min using the Ekblom Bak submaximal ergometer test
Change in motivation level | Change between baseline and 1-year follow-up
  Motivation to make lifestyle changes to improve health on an 11-point numerical rating scale.
Proportion achieved goals | Measured only at 1-year follow-up
  Proportion of goals achieved of the goals set by the intervention group at baseline
Change in fitness level | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for fitness where points are given for grade of deviation from norm. Minimum -2, maximum +2. Higher scores indicate better fitness level.
Change in strength upper extremity | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for strength upper extremity where points are given for grade of deviation from norm. Minimum -2, maximum +2. Higher scores indicate better strength.
Change in strength lower extremity | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for strength lower extremity where points are given for grade of deviation from norm. Minimum -2, maximum +2. Higher scores indicate better strength.
Change in strength trunk muscles | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for strength trunk where points are given for grade of deviation from norm. Minimum -2, maximum +2. Higher scores indicate better strength.
Change in balance | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for balance where points are given for grade of deviation from norm. Minimum -2, maximum +2. Higher scores indicate better balance.
Change in mobility | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for mobility where points are given for grade of deviation from norm. Minimum -2, maximum 0. Lower score indicates mobility dysfunction, 0 indicates normal mobility.
Change in posture | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for posture where points are given for grade of deviation from norm. Minimum -1, maximum 0. Lower score indicates postural deviations, 0 indicates normal postural measurements.
Change in weight measures | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for weight where points are given for grade of deviation from recommended values. Minimum -2, maximum 0. Lower score indicates overweight (or underweight), 0 indicates normal weight.
Change in pain | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for pain where points are given for number of pain locations, score on the Örebro Musculoskeletal Pain Screening Questionnaire and on the pain question on Euroqol-5 dimensions-3 levels. Minimum -2, maximum 0. Lower score indicates more pain, 0 indicates no pain.
Change in physical activity | Change between baseline and 1-year follow-up
  Point level on the study-specific functional profile arm for physical activity where points are given for grade of deviation from recommended values when objectively measured with accelerometers. Minimum -2, maximum +2. Increased point value indicates higher physical activity level.
Change in handgrip strength | Change between baseline and 1-year follow-up
  Measured with Jamar handdynamometer (kg)
Change in biceps strength | Change between baseline and 1-year follow-up
  Measured with 30-second biceps test (number repetitions)
Change in leg strength | Change between baseline and 1-year follow-up
  Measured with 30-second chair-stand test (number repetitions)
Change in calf strength | Change between baseline and 1-year follow-up
  Measured with single-foot heel rises (number repetitions)
Change in ventral trunk strength | Change between baseline and 1-year follow-up
  Measured with plank test (seconds)
Change in dorsal trunk strength | Change between baseline and 1-year follow-up
  Measured with back endurance test (seconds)
Change in lower trunk strength | Change between baseline and 1-year follow-up
  Measured with supine bridge test (seconds)
Change in static balance - 1 | Change between baseline and 1-year follow-up
  Measured with stand-on-one-leg-eyes-open test (seconds)
Change in static balance - 2 | Change between baseline and 1-year follow-up
  Measured with stand-on-one-leg-eyes-closed test (seconds)
Change in static balance - 3 | Change between baseline and 1-year follow-up
  Measured with sharpened Romberg test (seconds)
Change in dynamic balance | Change between baseline and 1-year follow-up
  Measured with functional reach test (centimeters)
Change in mobility - 1 | Change between baseline and 1-year follow-up
  Measured with sit-rise test (points)
Change in mobility - 2 | Change between baseline and 1-year follow-up
  Measured with finger-floor test (centimeters)
Change in mobility - 3 | Change between baseline and 1-year follow-up
  Measured with lateral flexion test (centimeters)
Change in hypermobility score | Change between baseline and 1-year follow-up
  Measured with Beighton hypermobility score with point values between 0 and 9 where score over 4 indicate general hypermobility.
Change in neck mobility | Change between baseline and 1-year follow-up
  Measured with occiput-to-wall test (points)
Change in foot pronation | Change between baseline and 1-year follow-up
  Measured with navicular drop test (millimeters)
Change in habitual stance | Change between baseline and 1-year follow-up
  Measured with patella mobility test (points)
Change in health-related quality of life assessed with EQ5D index | Change between baseline and 1-year follow-up
  Measured with index values for Euroqol-5 dimensions-3 levels. Minimum -0.59, maximum +1. Higher scores indicate better health-related quality of life.
Change in health-related quality of life assessed with EQ5D VAS | Change between baseline and 1-year follow-up
  Measured with the 100-point barometer for Euroqol-5 dimensions-3 levels. Minimum 0, maximum 100. Higher scores indicate better health-related quality of life.
Change in self-reported physical activity assessed with Swedish questionnaire | Change between baseline and 1-year follow-up
  Measured with Swedish National Board of Health and Welfare questionnaire with 2 questions on physical activity and exercise measured in minutes. Minimum 0, maximum measured value 540. Increasing values indicate higher levels of physical activity.
Change in self-reported physical activity assessed with Saltin Grimby Physical Activity Level Scale (SGPALS) | Change between baseline and 1-year follow-up
  Measured with SGPALS with point values between 1 and 4 where increasing values indicate higher level of physical activity.
Change in self-reported sedentary time | Change between baseline and 1-year follow-up
  Measured in hours per day with SED-GIH questionnaire with values between 0 and 24 where increasing sedentary time is considered to have a negative impact on health.
Change in risk for chronic pain and sickness absence assessed with Örebro Musculoskeletal Pain Screening Questionnaire | Change between baseline and 1-year follow-up
  Measured with Örebro Musculoskeletal Pain Screening Questionnaire with scores between 1 and 100 where increasing values indicate higher risk for chronic pain and sickness absence.
Change in number of pain locations | Change between baseline and 1-year follow-up
  Measured with a pain diagram
Change in proportion smokers | Change between baseline and 1-year follow-up
  Proportion smokers in each group
Change in proportion acceptable level blood glucose | Change between baseline and 1-year follow-up
  Proportion with blood glucose levels within recommended limits (4.0-6.0 mmol/L)
Change in proportion acceptable level serum cholesterol | Change between baseline and 1-year follow-up
  Proportion with cholesterol levels within recommended limits (3.3-6.9 mmol/L)
Change in proportion acceptable level triglycerides | Change between baseline and 1-year follow-up
  Proportion with triglyceride levels within recommended limits (0,45-2.6)
Change in proportion acceptable blood pressure | Change between baseline and 1-year follow-up
  Proportion of participants with blood pressure within recommended limits
Change in proportion normal body mass index (BMI) | Change between baseline and 1-year follow-up
  Proportion of participants with BMI within recommended limits
Change in proportion acceptable waist circumference | Change between baseline and 1-year follow-up
  Proportion of participants with waist circumference below recommended level
Change in stress symptoms assessed with Stress and Crisis Inventory-93 | Change between baseline and 1-year follow-up
  Measured with Stress and Crisis Inventory-93 questionnaire. Minimum 0, maximum 140, with higher values indicating higher stress levels.
Change in depression and anxiety symptoms assessed with Hospital Anxiety and Depression Scale | Change between baseline and 1-year follow-up
  Measured with Hospital Anxiety and Depression Scale. Minimum 0, maximum 42 with 21 as maximum for anxiety and 21 maximum for depression. Increasing values indicate more severe symptoms.
Correlation between self-assessed and objectively measured fitness | Change between baseline and 1-year follow-up
  Correlation between fitness self-assessed on a 5-point Likert scale and point value on the fitness arm on the study-specific functional profile. Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Correlation between self-assessed and objectively measured fitness - 2 | Change between baseline and 1-year follow-up
  Correlation between fitness self-assessed on a 5-point Likert scale and fitness grade on the Ekblom Bak fitness test (5 point Likert scale). Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Correlation between self-assessed and objectively measured strength upper extremity | Change between baseline and 1-year follow-up
  Correlation between upper extremity strength self-assessed on a 5-point Likert scale and point value for the strength upper extremity arm on the study-specific functional profile. Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Correlation between self-assessed and objectively measured strength lower extremity | Change between baseline and 1-year follow-up
  Correlation between lower extremity strength self-assessed on a 5-point Likert scale and point value for the strength lower extremity arm on the study-specific functional profile. Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Correlation between self-assessed and objectively measured balance | Change between baseline and 1-year follow-up
  Correlation between balance self-assessed on a 5-point Likert scale and point value on the balance arm on the study-specific functional profile. Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Correlation between self-assessed and objectively measured physical activity | Change between baseline and 1-year follow-up
  Correlation between self-assessed walking ability on a 5-point Likert scale and point value on the physical activity arm on the study-specific functional profile. Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Correlation between self-assessed and objectively measured physical activity - 2 | Change between baseline and 1-year follow-up
  Correlation between self-assessed walking ability on a 5-point Likert scale and number of daily minutes in moderate-to-very vigorous physical activity measured with accelerometers. Minimum -1, maximum +1. Higher values indicate better correlation between the 2 measures.
Change in relative physical activity | Change between baseline and 1-year follow-up
  Mean daily minutes of moderate-to-very vigorous physical activity measured with accelerometers for 1 week where moderate is individually calculated in relation to fitness level (46% of VO2max).
Change in sufficient physical activity | Change between baseline and 1-year follow-up
  Number of mean daily minutes of physical activity measured with accelerometers for 1 week above a known health-promoting level based on a fitness level of 31.5 ml/kg for women and 35 ml/kg for men.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Bornhöft, PhD, Principal Investigator — Region Västra Götaland, University of Gothenburg
Locations (1):
- Familjeläkarna i Mölnlycke, Mölnlycke, Region Västra Götaland, Sweden

IPD SHARING:
Plan to Share IPD: No